CLINICAL TRIAL: NCT02729844
Title: Pulmonary Hypertension in Preterm Children Born at Gestational Age <30 Weeks: Prevalence, Risk Factors and Outcome
Brief Title: Neolifes Heart - Pulmonary Hypertension in Preterm Children
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. R.M.F. Berger, Prof. Dr. R.M.F. Berger, University Medical Center Groningen
Other Study IDs: 201500715
Record Dates: First submitted 2016-03-21; First posted 2016-04-06 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Hypertension; Bronchopulmonary Dysplasia
Keywords: Incidence; Risk factors; Outcome
MeSH Terms: conditions — Hypertension, Pulmonary; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neolifes Heart: All premature infants, admitted at the neonatal intensive care unit (NICU) of the University Medical Centre Groningen, born <30 weeks or birth weight < 1000 gram, who participate in NeolifeS

SUMMARY:
NeoLifeS is a cohort follow up study that prospectively collects data of regular care of children born preterm in the University Medical Center Groningen (UMCG) and aims to improve the quality of care for these children.

NeoLifeS-Heart is a sub-study that focuses on the problem that a high proportion of preterm infants develop cardiovascular disorders. Related to the immaturity of their lungs, preterm infants are at risk to develop the condition Bronchopulmonary dysplasia (BPD). Also, the vasculature of the lungs is often not fully developed, making them more vulnerable for the development of Pulmonary Hypertension (PH), a high blood pressure in the lungs. 15-20% of the infants with extremely low birth weight are believed to develop PH, this proportion has been suggested to raise to 50% in infants with severe BPD. The presence of PH significantly worsens the prognosis and survival of these children.

The condition PH is insufficiently characterized. Knowledge of incidence, prevalence, risk factors for the development of PH and survival, will be the first step in improving detection strategies, possible treatment options and thereby prognosis and survival of these children.

Objective: To determine the incidence and prevalence of PH in preterm infants. In addition we aim to identify risk factors for the development of PH and determine the survival and prognosis of these preterm infants.

Study design: A prospective cohort study. Study population: All preterm infants, admitted at the neonatology UMCG, born <30 weeks and/or birth weight < 1000 gram, who participate in NeoLifeS Primary parameters: The occurrence of PH (Incidence and Prevalence).

Secondary parameters:

* Maternal and neonatal patient characteristics that are potential risk factors for the development of PH,
* Morbidity-score (quality of life and hospital admissions) and mortality.

DETAILED DESCRIPTION:
Background:

The development is not complete in premature born children. For example, the lungs are not fully developed. This is associated with shortness of breath and an increased oxygen need. Some of these children will need ventilation support and develop the condition Bronchopulmonary dysplasia (BPD). BPD is considered with lung injury and more than 28 days of ventilation support. These children have more need for oxygen and are extra sensitive for infections. In the present era, BPD most often occurs in extremely premature infants born at 24-28 weeks' post menstrual age, who have showed less severe acute respiratory symptoms and require less respiratory support than BPD patients have traditionally had in the past. Histological examination of these 'new BPD' patients suggests that the extreme preterm birth in combination with perinatal lung injury affects the normal growth of the lung development, resulting in disrupted vascular growth and impaired alveolarization, which could result in PH, a high blood pressure in the lungs. The causal relation among prenatal factors, prematurity, BPD and PH are not fully known yet. In premature newborns, < 30 weeks, the prevalence of BPD has been estimated to be 30-60% , while the prevalence of occurrence of PH received significantly less attention and estimates vary from 18% in the total group and up to 30% in the BPD-group and 50% in the severe BPD-group. The development of PH complicates the postnatal course of extreme premature infants. Both early and late PH are associated with poor outcomes among preterm infants, with and without BPD. Recent reports suggests that morbidity and late mortality of PH in the 'new BPD' is high, with up to 48% mortality 2 years after diagnosis of PH. The pathogenesis of BPD is complex and known risk factors for the development of severe BPD includes maternal and neonatal factors, such as childbearing history, male gender, smoking mother during pregnancy, chorioamnionitis, low-birth-weight, gestational age, cholestasis and acute lung injury by high ventilator settings. Risk factors for the development of PH in extreme preterm infants are not well defined. Knowledge of prevalence and risk factors of PH in extreme premature infants will allow evidence-based screening guidelines for the infants. Also potentially leading to prevention of this complicating condition in the future, since an earlier intervention will be possible under guidance of known risk factors. Early detection will lead to early and thus potentially better treatment of PH in preterm born infants.

Objective of the study:

Primary:

To identify the incidence and prevalence of PH in premature born infants with and without BPD in the first year of life.

Secondary:

To identify risk factors for the development of PH in these patients To characterize morbidity and survival of these patients during the first 2 yrs of life.

Study design:

Prospective Observational Cohort study. Inclusion 2016-2018, Follow up for standardized care (including QoL) at: 6, 12 and 24 months corrected age.

For Neolifes-Heart: echocardiography and transcutaneous oxygen measurement will be performed at: 1) first week after birth, 2) 3 months corrected age, 3) 12 months corrected age.

Study population:

All premature infants, admitted at the neonatology UMCG, born <30 weeks or birth weight < 1000 gram, who participate in NeolifeS. Only children whom parents have given written informed consent are included in this study.

Primary study parameter:

The echocardiographic presence of PH (incidence and point-prevalence).

Secondary study parameters:

Morbidity, Mortality: Quality of life questionnaire and survival. Maternal factors: mode of conception, delivery, preterm premature rupture of membranes (PROM), maternal disease history, illnesses during gestation, tabacco and medication use. Perinatal variables: slow growth patterns in utero, prenatal echo findings, PROM, chorioamnionitis, oligohydramnios, birth events, placental histology. Neonatal variables: development of BPD, low birth weight, gestational age, skull circumference, pulmonary and artificial ventilation variables, oxygen need, presence of persistent arterial duct (PDA), medication, infections, renal function, complications (NEC), slow growth at gestational age (GA) 36wks and at discharge. other: demographics, slow growth, admissions, medication, feeding, neurological development, respiratory symptoms, lung clearing index.

ELIGIBILITY:
Inclusion Criteria:

* All premature infants born <30 weeks or <100 gram
* admitted at the neonatology UMCG,
* participation in the study Neolifes

Exclusion Criteria:

* no informed consent

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All premature infants, admitted at the neonatology UMCG, born <30 weeks or birth weight < 1000 gram, who participate in NeolifeS
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of pulmonary hypertension | at 12 months corrected age.

SECONDARY OUTCOMES:
Mortality | At 12 months corrected age.
  survival
Morbidity | at 12 months corrected age
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Berger, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only in case of clinical need, the data of the echocardiograph will be available.

REFERENCES:
- [Background] Northway WH Jr, Rosan RC, Porter DY. Pulmonary disease following respirator therapy of hyaline-membrane disease. Bronchopulmonary dysplasia. N Engl J Med. 1967 Feb 16;276(7):357-68. doi: 10.1056/NEJM196702162760701. No abstract available. PMID 5334613
- [Background] Bancalari E, Claure N. Definitions and diagnostic criteria for bronchopulmonary dysplasia. Semin Perinatol. 2006 Aug;30(4):164-70. doi: 10.1053/j.semperi.2006.05.002. PMID 16860155
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Mourani PM, Sontag MK, Younoszai A, Miller JI, Kinsella JP, Baker CD, Poindexter BB, Ingram DA, Abman SH. Early pulmonary vascular disease in preterm infants at risk for bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2015 Jan 1;191(1):87-95. doi: 10.1164/rccm.201409-1594OC. PMID 25389562
- [Background] Berger RM, Beghetti M, Humpl T, Raskob GE, Ivy DD, Jing ZC, Bonnet D, Schulze-Neick I, Barst RJ. Clinical features of paediatric pulmonary hypertension: a registry study. Lancet. 2012 Feb 11;379(9815):537-46. doi: 10.1016/S0140-6736(11)61621-8. Epub 2012 Jan 11. PMID 22240409
- [Background] Khemani E, McElhinney DB, Rhein L, Andrade O, Lacro RV, Thomas KC, Mullen MP. Pulmonary artery hypertension in formerly premature infants with bronchopulmonary dysplasia: clinical features and outcomes in the surfactant era. Pediatrics. 2007 Dec;120(6):1260-9. doi: 10.1542/peds.2007-0971. PMID 18055675
- [Background] Bhat R, Salas AA, Foster C, Carlo WA, Ambalavanan N. Prospective analysis of pulmonary hypertension in extremely low birth weight infants. Pediatrics. 2012 Mar;129(3):e682-9. doi: 10.1542/peds.2011-1827. Epub 2012 Feb 6. PMID 22311993
- [Background] Mourani PM, Abman SH. Pulmonary vascular disease in bronchopulmonary dysplasia: pulmonary hypertension and beyond. Curr Opin Pediatr. 2013 Jun;25(3):329-37. doi: 10.1097/MOP.0b013e328360a3f6. PMID 23615175
- [Background] Van Marter LJ. Epidemiology of bronchopulmonary dysplasia. Semin Fetal Neonatal Med. 2009 Dec;14(6):358-66. doi: 10.1016/j.siny.2009.08.007. Epub 2009 Sep 26. PMID 19783238
- [Background] Roofthooft MT, Elema A, Bergman KA, Berger RM. Patient characteristics in persistent pulmonary hypertension of the newborn. Pulm Med. 2011;2011:858154. doi: 10.1155/2011/858154. Epub 2011 May 24. PMID 21660250
- [Background] Hilgendorff A, Reiss I, Ehrhardt H, Eickelberg O, Alvira CM. Chronic lung disease in the preterm infant. Lessons learned from animal models. Am J Respir Cell Mol Biol. 2014 Feb;50(2):233-45. doi: 10.1165/rcmb.2013-0014TR. PMID 24024524
- [Background] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- [Background] Ploegstra MJ, Roofthooft MT, Douwes JM, Bartelds B, Elzenga NJ, van de Weerd D, Hillege HL, Berger RM. Echocardiography in pediatric pulmonary arterial hypertension: early study on assessing disease severity and predicting outcome. Circ Cardiovasc Imaging. 2014 Dec 31;8(1):e000878. doi: 10.1161/CIRCIMAGING.113.000878. Print 2015 Jan. PMID 25552488